CLINICAL TRIAL: NCT05487352
Title: Diagnostic Efficiency Analysis of Oral Glucose Tolerance Test and Prediction Model Establishment in the First Trimester for Gestational Diabetes Mellitus: a Prospective Cohort Study
Brief Title: Diagnostic Analysis of Oral Glucose Tolerance Test in Early Pregnancy for Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20210134-R
Record Dates: First submitted 2022-07-21; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: gestational diabetes mellitus; first trimester; prediction model
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood was collected from subjects and divided into plasma and blood cells by centrifugation for preservation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hyperglycemia in the first trimester: The 75g oral glucose tolerance test was performed before 14 weeks of gestation, and any of the fasting, 1-hour and 2-hours blood glucose was ≥ 5.1, 10.0 and 8.5 mmol/L, respectively.
  Interventions: Other: hyperglycemia exposure in the first trimester
- euglycemia in the first trimester: The 75g oral glucose tolerance test was performed before 14 weeks of gestation, and the fasting, 1-hour and 2-hours blood glucose were all < 5.1, 10.0 and 8.5 mmol/L, respectively.

INTERVENTIONS:
Other: hyperglycemia exposure in the first trimester — The exposure means the hyperglycemia identified by the 75g oral glucose tolerance test before the 14 weeks of gestation
  Groups: hyperglycemia in the first trimester

SUMMARY:
The aim of this study is to explore the diagnostic efficacy of oral glucose tolerance test in early pregnancy and establish the prediction model for gestational diabetes mellitus, so as to provide the optimal screening of gestational diabetes mellitus in the first trimester. The treatment started when the pregnancy was confirmed by transvaginal ultrasound (around 6 weeks of gestation) and continued until 42 days postpartum. The study is a single center, prospective cohort study. A total of 781 participants within 14 weeks of gestation were recruited.

ELIGIBILITY:
Inclusion Criteria:

* 1. Intrauterine pregnancy within 7-14 weeks of gestation
* 2. 20-45 years of age
* 3. Singleton pregnancy
* 4. Giving informed consent and willing to participate in this study
* 5. Planning to give birth in Women's Hospital School of Medicine Zhejiang University

Exclusion Criteria:

* 1. Pre-existing diabetes
* 2. Taking medications that may affect blood glucose levels within one month
* 3. Participating in other intervention studies
* 4. Recurrent abortion, threatened abortion, cervical incompetence or fetal malformation

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Subjects were confirmed "intrauterine live birth" by ultrasound examination and were during 7-14 weeks of gestation confirmed by the combination of their last menstrual period and nuchal translucency ultrasound examination.
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
gestational diabetes mellitus | 24-28 weeks of gestation
  any of the fasting, 1-hour and 2-hour blood glucose ≥ 5.1, 10.0, 8.5 mmol/L, respectively, in the 75g oral glucose tolerance test during 24-28 weeks of gestation

SECONDARY OUTCOMES:
gestational weight gain | before delivery
  total weight gain from pre-pregnancy until delivery
gestational age at delivery | through study completion, an average of 39 gestational weeks
  gestational weeks at the day of delivery
birthweight | within 24 hours after birth
  birthweight of the infant
neonatal weight, height and head circumference | 42 days after birth
  baby's weight, height and head circumference at 42 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhang, Dr, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association Professional Practice Committee. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S17-S38. doi: 10.2337/dc22-S002. PMID 34964875
- [Background] Wang H, Li N, Chivese T, Werfalli M, Sun H, Yuen L, Hoegfeldt CA, Elise Powe C, Immanuel J, Karuranga S, Divakar H, Levitt N, Li C, Simmons D, Yang X; IDF Diabetes Atlas Committee Hyperglycaemia in Pregnancy Special Interest Group. IDF Diabetes Atlas: Estimation of Global and Regional Gestational Diabetes Mellitus Prevalence for 2021 by International Association of Diabetes in Pregnancy Study Group's Criteria. Diabetes Res Clin Pract. 2022 Jan;183:109050. doi: 10.1016/j.diabres.2021.109050. Epub 2021 Dec 6. PMID 34883186
- [Background] Saravanan P; Diabetes in Pregnancy Working Group; Maternal Medicine Clinical Study Group; Royal College of Obstetricians and Gynaecologists, UK. Gestational diabetes: opportunities for improving maternal and child health. Lancet Diabetes Endocrinol. 2020 Sep;8(9):793-800. doi: 10.1016/S2213-8587(20)30161-3. Epub 2020 Aug 18. PMID 32822601
- [Background] McIntyre HD, Catalano P, Zhang C, Desoye G, Mathiesen ER, Damm P. Gestational diabetes mellitus. Nat Rev Dis Primers. 2019 Jul 11;5(1):47. doi: 10.1038/s41572-019-0098-8. PMID 31296866
- [Background] Catalano PM, McIntyre HD, Cruickshank JK, McCance DR, Dyer AR, Metzger BE, Lowe LP, Trimble ER, Coustan DR, Hadden DR, Persson B, Hod M, Oats JJ; HAPO Study Cooperative Research Group. The hyperglycemia and adverse pregnancy outcome study: associations of GDM and obesity with pregnancy outcomes. Diabetes Care. 2012 Apr;35(4):780-6. doi: 10.2337/dc11-1790. Epub 2012 Feb 22. PMID 22357187
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375